CLINICAL TRIAL: NCT03307551
Title: Evaluation of Automated Delivery of Propofol Using Closed-Loop Anaesthesia Delivery System in Patients Undergoing Thoracic Surgery: A Randomised Controlled Study
Brief Title: Evaluation of Automated Propofol Delivery in Patients Undergoing Thoracic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Nitin Sethi (Other)
Responsible Party: Sponsor-Investigator, Dr Nitin Sethi, Associate Professor & Consultant, Sir Ganga Ram Hospital
Organization: Sir Ganga Ram Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EC/09/17/1254
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Thoracic Diseases; Surgery
Keywords: propofol, automated, manual
MeSH Terms: conditions — Thoracic Diseases | interventions — Propofol

STUDY DESIGN:
Intervention Model Description: 30-patients aged 18-65 years, ASA physical status I-III, of either sex, and undergoing unilateral open thoracic surgery or unilateral video-assisted thoracic surgery (VATS) will randomly allocated by computer generated numbers to one of the following two groups of 15 patients each:
  Group-1 [CLADS Group, n=15, Study group]: Anaesthesia will be induced and maintained with propofol administered using the automated CLADS.
  Group-2 [Manual Group, n=15, Control group]: Anaesthesia will be induced and maintained with propofol administered using manually controlled infusion pumps titrated to BIS scores.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded to the type of anaesthesia intervention.The attending anaesthesiologist will however not be blinded to the technique utilized to administer GA and recovery immediately after extubation inside the OR. The postoperative patient recovery profile will be evaluated by an independent assessor blinded to the technique of GA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CLADS group (Active Comparator): Anaesthesia will be induced and maintained with Propofol administered by CLADS. Its administration rate will be controlled by a feedback loop facilitated by BIS monitoring. A BIS value of 50 will be used as the target point for induction and maintenance of anaesthesia.
  Interventions: Drug: Propofol
- Manual group (Active Comparator): Anaesthesia will be induced and maintained with propofol administration by an intravenous infusion pump. Its administration rate will be controlled manually to maintain a target BIS of 50 during induction and maintenance of anaesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol delivery will be controlled using automated closed loop anaesthesia delivery system which will control propofol delivery rate to consistent anaesthetic depth (BIS-50) feedback from the patient (CLADS group)
  Arms: CLADS group
Drug: Propofol — Propofol delivery will be controlled using infusion pumps which will be manually controlled to deliver propofol to maintain consistent anaesthetic depth (BIS-50). (Manual group)
  Arms: Manual group

SUMMARY:
Automated delivery of propofol using computer-controlled closed loop anaesthesia device delivers propofol based on patient's frontal cortex electrical activity as determined by bi-spectral index (BIS). Evaluation of anaesthesia delivery by these systems has shown that they deliver propofol and maintain depth of anaesthesia with far more precision as compared to manual administration.

By automatically controlling anaesthesia depth consistency they provide time to the anaesthesiologist to focus on other aspects of patient care such as managing intra-operative hemodynamics and ventilation perturbations during major surgeries.

Closed loop anaesthesia delivery system (CLADS) is an indigenously developed continuous automated intravenous infusion system which delivers propofol based on patients EEG profile (BIS) feedback. Although a few studies have already evaluated these automated systems in patients undergoing thoracic surgery, but suffered from significant limitations (small number of patients, not dedicated to thoracic surgery cohort). Currently, there is no data available regarding CLADS performance vis a vis adequacy of GA and haemodynamic profile in patients undergoing thoracic surgery.

We contend that propofol as delivered by CLADS will proffer greater consistency to anaesthesia depth, intra-operative hemodynamic stability, and rapid recovery upon anaesthesia discontinuation than manual means of delivering propofol TIVA. This randomised controlled study aims to compare the efficiency of CLADS-driven propofol TIVA versus manually controlled propofol TIVA in patients undergoing thoracic surgery.

DETAILED DESCRIPTION:
After Ethics Committee approval and written informed consent, thirty-participants (30 per group) aged 18-65 years, ASA physical status I-III, of either sex, and undergoing unilateral open thoracic surgery or unilateral video-assisted thoracic surgery (VATS) will be included in this single centre (Sir Ganga Ram Hospital, New Delhi-110060, India) prospective, single-blinded, two-arm, randomised controlled study.

The patients who qualify inclusion criteria and consent for recruitment will be randomly divided into one of the two groups:

Group-1 [CLADS Group, n=15, Study group]: Anaesthesia will be induced and maintained with propofol administered using the automated CLADS.

Group-2 [Manual Group, n=15, Control group]: Anaesthesia will be induced and maintained with propofol administered using manually controlled infusion pumps titrated to BIS scores.

Sample-size Estimation In a previous multi-centre study, the percentage of time the BIS was within 10 percentage of the target BIS was 81.4 percent in the CLADS group versus 55.34 percent in the manual group. Based on the above, to detect 20 percent difference in the two groups, a sample size of 12 patients per group to provide 90 percent power with a bilateral alpha risk value of 0.05 will be required. We plan to recruit a total of 30 patients to cover up for unanticipated losses after the recruitment.

Randomisation, Allocation Concealment The patients will be randomly allocated to one of the two groups based on a computer-generated random number table. Randomisation sequence concealment will include opaque-sealed envelopes with alphabetic codes whose distribution will be in control of an independent analyst. The envelopes will be opened; patient's data-slip will be pasted on them, and will be sent back to the control analyst.

Blinding Strategy Inside the OR, the attending anaesthesiologist will not be blinded to the technique utilised to administer GA and the recovery parameters immediately after extubation. However, the postoperative patient recovery profile will be evaluated by an independent assessor blinded to the GA technique and periextubation profile.

Management of Anesthesia Two peripheral venous lines (18G/20G catheter) will be secured. Invasive vascular access (arterial line for direct continuous blood pressure assessment, central venous catheter) will be secured as per the requirement of surgery. Standard monitoring (EKG, NIBP, pulse oximeter, EtCO2) will be applied. A BIS sensor (Covidien IIc, Mansfield, USA) will be applied over the patient's forehead according to manufacturer's instructions (Model DSC-XP, Aspect medical system, USA) prior to induction of anaesthesia for continuous monitoring of depth-of-anaesthesia.

Anaesthesia Technique

All the patients will receive pre-induction fentanyl-citrate 2 mcg/kg and anesthesia will be induced with propofol. In the CLADS group, propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring. A BIS value of 50 will be used as the target point for induction and maintenance of anesthesia. The Manual group would comprise manual propofol administration by an intravenous infusion pump to maintain a target BIS of 50 during induction and maintenance of anesthesia.

After induction of anesthesia, atracurium besylate 0.05mg/kg will be given to facilitate tracheal intubation. In order to facilitate one lung ventilation (OLV) patients trachea will be intubated using appropriate-sized double-lumen tube in all the patients. Oxygen-air mixture (FiO2 0.50) will be used for intraoperative ventilation in both the groups. In addition, starting the period after tracheal intubation, all the patients will receive 1 mcg/kg/hr fentanyl infusion for intraoperative analgesia. Intraoperative muscle relaxation will be maintained using atracurium infusion controlled by train-of-four response on peripheral neuromuscular monitor (Infinity TridentNMT Smartpod, Draeger Medical Systems, Inc Telford, USA).

In all patients undergoing open thoracic surgery, a thoracic epidural catheter will be placed in the indicated intervertebral space for facilitating postoperative analgesia.

Thirty minutes before the end of surgery, non-opioid analgesics, such as paracetamol 1-gm, tramadol 100 mg and/or diclofenac 75 mg will be administered to all the patients. Propofol delivery will be stopped at the point of completion of skin closure. Residual neuromuscular blockade (assessed with train-of-four response) will be reversed with neostigmine (50 µg/kg) and glycopyrrolate (20 µg/kg). Tracheal extubation will be undertaken if planned post-extubation ventilation is not instituted and the patients are wide awake and obeying commands.

Assessment Parameters Intraoperative

1. Adequacy of anaesthesia depth will be determined by the percentage of the valid CLADS time during which the BIS remained within 10% of the target BIS (50), median absolute performance error (MDAPE), wobble and global score (Varvel criteria)
2. Haemodynamic parameters such a heart rate, non-invasive blood pressure will be recorded
3. Early recovery from anaesthesia profile which includes time to eye opening and time to extubation after discontinuation of anesthesia will be noted

Postoperative

1. Sedation will be assessed using Modified Observer's assessment of alertness/sedation scale.
2. Incidence of awareness will be determined using Modified Brice Questionnaire.

After discontinuation of anaesthesia delivery (0-time point) the time to eye opening and time to extubation will be determined. After tracheal extubation, the patients will be shifted to postoperative recovery room adjoining OT suites and will be closely observed for oxygenation and ventilation status, pain (numeric rating score) and sedation. Patients with epidural catheter in-situ will be started with PCEA pump for pain relief. Patients will be analysed for intra-operative awareness using Modified Brice Questionnaire (24 hours, 48 hours postoperatively).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* undergoing unilateral open thoracic surgery or unilateral video-assisted thoracic surgery (VATS) Exclusion Criteria:

Exclusion Criteria:

* Uncompensated cardiovascular disease (e.g. uncontrolled hypertension, atrio-ventricular block, sinus bradycardia, congenital heart disease, reduced LV compliance, diastolic dysfunction)
* Hepato-renal insufficiency
* Uncontrolled endocrinology disease (e.g. diabetes mellitus, hypothyroidism)
* Known allergy/hypersensitivity to the study drug
* Drug dependence/substance abuse
* Requirement of postoperative ventilation
* Refusal to informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Anaesthesia depth consistency using BIS scores | From beginning of anaesthesia (0-hours, baseline) till 10 hours intraoperatively
  Determined by the percentage of the total anaesthesia time in which the BIS scores remain within a score of 10% of the target BIS (i.e. BIS-50) in both the study arms.

SECONDARY OUTCOMES:
Performance Characteristic of propofol anaesthesia delivery system | From beginning of anaesthesia (0-hours, baseline) till 10 hours intraoperatively
  Determined by using Varvel criteria parameters; median performance error (MDP), median absolute performance error (MDAPE), wobble and global score in both the study arms
Change in Intra-operative heart Rate (beats per minute) | From beginning of anaesthesia (0-hours, baseline) till 10 hours intraoperatively
  Comparison of intra-operative heart rate between both the arms will be done
Change in Intra-operative systolic , diastolic, and mean (mmHg) | From beginning of anaesthesia (0-hours, baseline) till 10 hours intraoperatively
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean between both the arms will be done
Recovery from anesthesia | From end of anaesthesia till 20-minutes postoperatively]
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Recovery from anesthesia | From end of anaesthesia till 20-minutes postoperatively]
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Intra-operative awareness | From the end of anaesthesia till 48-hours postoperatively
  Will be assessed using modified brice questionnaire
Propofol induction dose (mg) | From start of propofol injection till 2- minutes intraoperatively
  Dose of propofol required for induction of anaesthesia
Propofol maintenance dose (mg/kg/hr) | From 2-minutes intraoperatively till 10-hours intraoperatively
  Dose of propofol required for maintenance of anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Goverdhan D Puri, MD, PhD, Study Chair — Post Graduate Institute of Medical Education & Research, Chandigarh, India; Jayashree Sood, MD,FFRCA, Study Director — Sir Ganga Ram Hospital
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No